CLINICAL TRIAL: NCT04029649
Title: The Role of Beta-1,3/1,6-D-Glucan From Mycelium Extract of Indonesian Ganoderma Lucidum on Ulcerative Colitis: A Double-Blind Randomized Controlled Trial
Brief Title: Beta-1,3/1,6-D-Glucan Ganoderma Lucidum on Ulcerative Colitis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fakultas Kedokteran Universitas Indonesia (Other)
Responsible Party: Principal Investigator, Marcellus Simadibrata, Prof. PhD., SpPD, KGEH, Professor, Fakultas Kedokteran Universitas Indonesia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19-01-0083
Record Dates: First submitted 2019-07-17; First posted 2019-07-23 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Ulcerative Colitis
Keywords: Beta-1,3/1,6-D-Glucan; Ganoderma lucidum; Ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beta-1,3/1,6-D-Glucan Ganoderma lucidum (Experimental): This group received capsule contains 180 mg Beta-1,3/1,6-D-Glucan from mycelium extract of Ganoderma lucidum with dose 3x1 capsule a day for 90 days
  Interventions: Drug: Beta-1,3/1,6-D-Glucan
- Placebo (Placebo Comparator): This group received empty capsule with dose 3x1 capsule a day for 90 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Beta-1,3/1,6-D-Glucan — Beta-1,3/1,6-D-Glucan capsule three times daily for 90 days
  Arms: Beta-1,3/1,6-D-Glucan Ganoderma lucidum
Drug: Placebo — Placebo capsule three times daily for 90 days
  Arms: Placebo

SUMMARY:
The aim of this study is to determine the efficacy and safety of Beta-1,3/1,6-D-Glucan from mycelium extract of Ganoderma lucidum on ulcerative colitis

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years old
* ulcerative colitis patients who are treated by 5-aminosalicylic acid (5-ASA) 3x500 mg
* agreed to participate in this study

Exclusion Criteria:

* ulcerative colitis patients who are treated by corticosteroid, immunosuppressive agents and biologic agents
* allergic to Ganoderma lucidum
* could not be randomised and participate in this study by clinical judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of Life: SF-36 questionnaire | 0 and 90 days
  Quality of Life is assessed by Indonesian validated Short Form 36 (SF-36) questionnaire. This questionnaire consist of 36 items/questions that evaluate quality of life in some elements. The elements are change in health (1 item), general health perception (5 items), energy/fatigue (4 items), mental health (5 items), social functioning (2 items), pain (2 items), physical functioning (10 items), role limitations due to emotional problems (3 items) and role limitations due to physical problems (4 items). The score from each question will be summed. Minimum score is 36 and maximum score is 138. Higher score indicates higher quality of life and lower score indicates lower quality of life. Higher score post intervention administration represents a positive outcome

SECONDARY OUTCOMES:
Change of C-Reactive Protein (CRP) level | 0 and 90 days
  Level of CRP is obtained from laboratory test.
Change of Erythrocyte Sedimentation Rate (ESR) | 0 and 90 days
  ESR is obtained from laboratory test.
Change of Tumor Necrosis Factor Alpha (TNF-α) level | 0 and 90 days
  Level of TNF-α is obtained from laboratory test
Change of Interleukin 6 (IL-6) level | 0 and 90 days
  Level of IL-6 is obtained from laboratory test
Change of fecal calprotectin level | 0 and 90 days
  Level of fecal calprotectin is obtained from stool examination
Change of Mayo score | 0 and 90 days
  Mayo score is assessed from colonoscopy. 0 = normal 1 = mild (erythema, decreased vascular pattern, mild friability) 2 = moderate (marked erythema, absent vascular pattern, friability, erosions) 3 = severe (spontaneous bleeding, ulceration)
Number of patients with neutrophils infiltrating crypt epithelium in colon biopsy | 0 and 90 days
  Colon biopsy is obtained from colonoscopy and histopathology examination

OTHER OUTCOMES:
Number of participants with adverse events (AEs) | 30, 60 and 90 days
  Number of participants with AE in this study
Number of participants with serious adverse events (SAEs) | 30, 60 and 90 days
  Number of participants with SAEs in this study

CONTACTS AND LOCATIONS:
Overall Officials: Marcellus Simadibrata, Principal Investigator — Division Of Gastroenterology Department Of Internal Medicine Faculty Of Medicine Universitas Indonesia
Locations (1):
- RSUPN dr. Cipto Mangunkusumo (Cipto Mangunkusumo Hospital), Jakarta, Jakarta Pusat, Indonesia

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-30): https://cdn.clinicaltrials.gov/large-docs/49/NCT04029649/Prot_SAP_002.pdf